CLINICAL TRIAL: NCT01675050
Title: A Placebo-controlled Crossover Trial Using Cyproheptadine To Treat Children With Functional Abdominal Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the wide availability of the drug in clinical practice, it was impossible to recruit adequate numbers for scientific power.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ismaeel Hashemi, Fellow Physician, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00056045
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Functional Abdominal Pain
MeSH Terms: interventions — Cyproheptadine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyproheptadine first then Placebo (Experimental): 4 weeks of cyproheptadine or placebo with crossover to the other
  Interventions: Drug: Cyproheptadine; Drug: sugar pill
- Sugar Pill first then Cyprotheptadine (Experimental): 4 weeks of cyproheptadine or placebo with crossover to the other
  Interventions: Drug: Cyproheptadine; Drug: sugar pill

INTERVENTIONS:
Drug: Cyproheptadine — 4 weeks of cyproheptadine or placebo with crossover to the other
  Other Names: Periactin
Drug: sugar pill — 4 weeks of cyproheptadine or placebo with crossover to the other
  Other Names: placebo

SUMMARY:
The investigators hypothesize that using Cyproheptadine in a placebo-controlled crossover trial would help relieve abdominal pain associated with (Functional Abdominal Pain (FAP) in children, achieving a greater response than that observed with placebo. In addition to assessing self-report of pain and other symptoms, the investigators also propose to perform experimental somatic pain testing to determine if there is evidence of peripherally-maintained central sensitization in children with FAP. The investigators also hypothesize that there will be an increase in somatic pain threshold after completion of a Cyproheptadine course compared to baseline testing prior to treatment, and compared to placebo. This would allow children with FAP to return to normal function, improve symptoms and overall general well-being

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 18 years-old
* Diagnosed with Functional Abdominal Pain using the Rome III Criteria must include all* of the following:

  1. Episodic or continuous abdominal pain
  2. Insufficient criteria for other FGIDs
  3. No evidence of an inflammatory, anatomic, metabolic, or neoplastic process that explains the subject's symptoms

     * Criteria fulfilled at least once per week for at least 2 months prior to diagnosis
* Written informed consent obtained from the patient/guardian before the initiation of any study-specific procedures

Exclusion Criteria:

* Age < 8 years-old or Age >18 years-old
* Child or parent are non-English speakers
* Child is using other CNS depressants (cyproheptadine causes drowsiness, and may enhance the adverse/toxic effect of other CNS Depressants e.g. opioids, barbiturates, Droperidol, Hydroxyzine, Alcohol)(29)
* Child has a history of hypersensitivity to Cyproheptadine products
* Child is currently using monoamine oxidase inhibitor (MAOI e.g. Nardil, Marplan, Parnate) (can cause a prolonged or intensified anticholinergic effect)
* Child was treated with Cyproheptadine in the past 4 weeks
* Child is currently using anticholinergic (can cause an additive anticholinergic effect e.g. Pramlintide)
* Concomitant SSRI use ( being a serotonin antagonist, may oppose effects)
* Concomitant use of Betahistine: Antihistamines may diminish the therapeutic effect of Betahistine
* Concomitant use of Acetylcholinesterase Inhibitors (Central): Anticholinergics may diminish the therapeutic effect of Acetylcholinesterase Inhibitors (Central) and vice versa.
* Child has a personal history of glaucoma
* Child has asthma (can cause thickening of bronchial secretions) (27,28)
* History of liver dysfunction/disease (can cause hepatitis)
* History of cardiac disease (not specific to Cyproheptadine, antihistamines have been associated with hypotension, palpitations, tachycardia and arrhythmias) (28,29).
* Females who are known to be pregnant will also be excluded. All females who are of child bearing age, or are already menstruating will perform a urine pregnancy test before enrolling.
* Any children who have difficulties swallowing tablets will receive teaching on how to swallow tablets. If they are still unable to do so, they will not participate in the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismaeel Hashemi, MD, Principal Investigator — University of Michigan
Locations (1):
- UmichiganHS, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyproheptadine First, Then Placebo: 4 weeks of cyproheptadine with crossover to 4 weeks of placebo.
- Sugar Pill First, Than Cyproheptadine: 4 weeks of placebo (sugar pill) with crossover to 4 weeks of cyproheptadine
Period: Period One Treatment
Arm/Group | Cyproheptadine First, Then Placebo | Sugar Pill First, Than Cyproheptadine
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Wash Out Period
Arm/Group | Cyproheptadine First, Then Placebo | Sugar Pill First, Than Cyproheptadine
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0
Period: Second Period Treatment
Arm/Group | Cyproheptadine First, Then Placebo | Sugar Pill First, Than Cyproheptadine
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cyproheptadine Then Placebo: 4 weeks of cyproheptadine with crossover to 4 weeks of placebo.
- Placebo Then Cyproheptadine: 4 weeks of placebo (sugar pill) with crossover to 4 weeks of cyproheptadine
- Total: Total of all reporting groups
Arm/Group | Cyproheptadine Then Placebo | Placebo Then Cyproheptadine | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 12.5 [9 to 16] | 10.5 [9 to 12] | 11.5 [9 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4
Pressure Pain Threshold [Mean (Standard Deviation); unit: kg/cm^2] — Increasing pressures are applied with a pressure plunger to the participants' thumbnail. The pressure at which the participant said that s/he felt pain is noted. The pressure is measured in in kilograms divided by centimeters squared. Population: Because 1 participant on the Cyproheptadine first side dropped out prior to assignment to placebo, there is only 1 participant shown on the cyproheptadine first then placebo side for the second baseline after washout prior to placebo.
  kg/cm^2
    Baseline prior to First Treatment | 1.75 (2) | 1.28 (.53) | 1.51 (.99)
    Baseline prior to Second Treatment: number analyzed (Participants) | 1 | 2 | 3
    Baseline prior to Second Treatment | 1.25 (0) | 1.08 (.18) | 1.13 (.16)
Improvement in Abdominal Pain [Mean (Standard Deviation); unit: units on a scale] — This is a pain scale derived from the abdominal pain Index child version, where on a scale of zero to 10, zero represents no pain, and ten represents the most pain possible Population: Because 1 participant in the Cyproheptadine first group withdrew prior to washout, that participant's data is not included in the pre-placebo period baseline.
  units on a scale
    Baseline prior to First Treatment | 4 (5.66) | 8.5 (2.12) | 6.25 (4.35)
    Baseline prior to Second Treatment: number analyzed (Participants) | 1 | 2 | 3
    Baseline prior to Second Treatment | 6 (0) | 6.5 (3.45) | 6.33 (2.52)

OUTCOME MEASURES:

1. Primary Outcome: Pressure Pain Threshold
Description: Increasing pressures were applied with a pressure plunger to the participants' thumbnail. The pressure at which the participant said that s/he felt pain is noted. The pressure is measured in kilograms by centimeters squared.
Time Frame: at 4 weeks of cyproheptadine or placebo treatment
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | All Participants Post Cyproheptadine | All Participants Post Placebo
Number analyzed (Participants) | 4 | 3
kg/cm^2 | 1.15 (.73) | 1.23 (.39)

2. Secondary Outcome: Abdominal Pain
Description: Participants rated the highest intensity of abdominal pain they experienced during the past two weeks on a scale of 0 (No Pain) to 10 (The Most Pain Possible), as derived from the "Abdominal Pain Index - Child Version" (Laird et al. 2015. Journal of Pediatric Psychology, 40(5), 517-525).
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants Post Cyproheptadine | All Participants Post Placebo
Number analyzed (Participants) | 4 | 3
units on a scale | 5.25 (4.11) | 8 (2)

ADVERSE EVENTS:
Time Frame: 10 weeks during study
Groups:
- Cyproheptadine: All participants while on Cyproheptadine.
- Placebo: All participants while on Placebo.
Arm/Group | Cyproheptadine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 3/4 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyproheptadine (N=4) | Placebo (N=3)
Increase Appetite (General disorders) | 1 | 1
Somnolence (Drowsiness) (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0
Cold Sweats (Vascular disorders) | 1 | 0
Restless Sleeping Pattern (Psychiatric disorders) | 1 | 0
Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Trouble Sleeping (Insomnia) (Psychiatric disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Statistical analyses were not conducted due to small sample size. Results should be interpreted with extreme caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes